CLINICAL TRIAL: NCT02399878
Title: Intra-operative Inspiratory Oxygen Fraction and Postoperative Respiratory Complications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, MD, PhD, Associate Professor, Massachusetts General Hospital
Other Study IDs: 03-2015
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Failure; Acute Respiratory Failure Requiring Intubation; Pulmonary Edema; Pneumonia; Surgical Wound Infection; Mortality
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Edema; Pneumonia; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing surgery: All non-cardiothoracic surgical patients aged 18 years or above receiving general anesthesia at Massachusetts General Hospital between January 2007 and August 2014.
  Interventions: Drug: Inspiratory oxygen

INTERVENTIONS:
Drug: Inspiratory oxygen

SUMMARY:
Respiratory complications represent the second most frequent type of postoperative complications with an incidence estimated to range from 2.0% to 7.9%

It has been shown that intra-operative protective ventilation is associated with a reduced risk of respiratory complications. The effects of intra-operative inspiratory oxygen fraction (FiO2) remain to be investigated.

In this study, the investigators aim to investigate the association between intra-operative FiO2 and respiratory complication as well as surgical site infection and ICU admission in patients undergoing non-cardiothoracic surgery. The investigators primary hypothesis is that high intra-operative FiO2 increases the risk of postoperative respiratory complications independent of predefined risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiothoracic surgery at Massachusetts General Hospital between January 2007 and August 2015
* Tracheally intubated at the beginning of the procedure and extubated at the end of the procedure
* above18 years of age

Exclusion Criteria:

* Missing information regarding main characteristics or the exposure variable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All non-cardiothoracic surgical patients aged 18 years or above receiving general anesthesia at Massachusetts General Hospital between January 2007 and August 2014
Sampling Method: Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2007-01; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Postoperative respiratory complications | 7 days after surgery

SECONDARY OUTCOMES:
Postoperative reintubation | 7 days after surgery
Postoperative respiratory failure | 7 days after surgery
Postoperative pneumonia | 7 days after surgery
Postoperative pulmonary edema | 7 days after surgery
Postoperative surgical site infection | 21 days after surgery
Postoperative admission to the intensive care unit | 7 days after surgery
Postoperative mortality | 7 days after surgery
Postoperative mortality | 30 days after surgery
Postoperative length of stay | 360 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — MGH

REFERENCES:
- [Derived] Staehr-Rye AK, Meyhoff CS, Scheffenbichler FT, Vidal Melo MF, Gatke MR, Walsh JL, Ladha KS, Grabitz SD, Nikolov MI, Kurth T, Rasmussen LS, Eikermann M. High intraoperative inspiratory oxygen fraction and risk of major respiratory complications. Br J Anaesth. 2017 Jul 1;119(1):140-149. doi: 10.1093/bja/aex128. PMID 28974067